CLINICAL TRIAL: NCT06569563
Title: Innervation Characteristics and Determination of Nerve Entry Points of the Musculus Semispinalis Capitis
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Seda GÖZENER CANBÜLBÜL, Principal Investigator, Medipol University
Other Study IDs: İMU-SEDAGOZENER-002
Record Dates: First submitted 2024-08-15; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Peripheral Nerve Disease; Muscular Injury
Keywords: m. semispinalis capitis; paraspinal muscle; muscle innervation mapping; cervical spine surgery; musculoskeletal anatomy; nerve entry point; intramuscular injection; cervical dystonia; botulinum toxin injections; innervation
MeSH Terms: conditions — Peripheral Nervous System Diseases; Torticollis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to determine the innervation characteristics and nerve entry points of the musculus semispinalis capitis. This muscle, which is involved in the extension of the head and neck, is a large and long cervico-thoracic muscle innervated by the dorsal rami of the cervical spinal nerves. The study seeks to enhance the effectiveness of procedures like electromyography (EMG) electrode placement and botulinum toxin injections used for diagnosing and treating conditions related to head and neck pain.

Accurately identifying these nerve entry points is crucial for ensuring the safety and efficacy of treatments, particularly for conditions like cervical dystonia and headaches. While existing studies have focused on the innervation and nerve mapping of various muscles, there has been no specific research on the nerve entry points of the musculus semispinalis capitis. This study aims to provide detailed knowledge of these aspects, offering valuable guidance for interventions in this area.

DETAILED DESCRIPTION:
The musculus semispinalis capitis, one of the cervical paraspinal muscles, originates from the transverse processes of the last cervical and the first six to seven thoracic vertebrae. It extends upward along both sides of the posterior midline and inserts between the superior and inferior nuchal lines on the occipital bone. This muscle is innervated by the dorsal rami of the cervical spinal nerves. As a large and long cervico-thoracic muscle, its primary function is the extension of the head and neck.

The aim of this study is to determine the innervation characteristics and nerve entry points of the musculus semispinalis capitis to enhance the effectiveness of procedures such as the placement of electromyography (EMG) electrodes for diagnostic and therapeutic purposes, as well as botulinum toxin injections used for treating conditions associated with head and neck pain.

The innervation characteristics and nerve entry points of the musculus semispinalis capitis need to be precisely identified, particularly in relation to treatments such as botulinum toxin injections for the management of spasms and pain in conditions like cervical dystonia, and for the treatment of headaches. Accurate identification of these points is crucial for ensuring safe and effective injections in this region and for understanding the anatomical variations in the area.

While there are studies in the literature focusing on the innervation characteristics and nerve entry points of various muscles, as well as nerve mapping, there has been no specific research on nerve entry point mapping for the musculus semispinalis capitis. Conducting this study will establish a detailed understanding of the innervation characteristics and nerve entry points of this muscle, providing valuable guidance for interventions in this area.

Previous studies on deep neck muscles have shown that procedures such as injections and EMG measurements have generally been performed using approximate localization methods. This study aims to use the results obtained to make these procedures more effective and less invasive.

ELIGIBILITY:
Inclusion Criteria:

* Cadavers were preserved using a 10% formalin solution.

Exclusion Criteria:

* neck and back region curvature,
* neck flexion and extension,
* related region muscle or nerve pathology,
* fracture,
* cadavers that have undergone previous surgery

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was conducted using 10 adult male cadavers, aged between 45 and 75 years, that had been fixed in 10% formalin solution. These cadavers were sourced from the laboratory of the Department of Anatomy at Ege University Faculty of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
The number of nerves innervating the semispinalis capitis muscle | 10 months
  The semispinalis capitis muscle is innervated by many nerves, primarily the dorsal branches of the cervical spinal nerves. The number of branches of the dorsal branches of the cervical nerves that enter the muscle was determined and counted one by one.
The location of nerves innervating the semispinalis capitis muscle | 10 months
  In order to determine which cervical nerve branch of the semispinalis capitis muscle was concentrated in which areas of the muscle, the perpendicular distances of the points where the nerves entered the muscle to the determined landmarks were measured and recorded in mm.
The thickness of nerves innervating the semispinalis capitis muscle | 10 months
  The thickness of the nerves innervating the semispinalis capitis muscle was measured and recorded.
Mapping of nerves innervating the semispinalis capitis muscle | 10 months
  After detailed information about the nerves innervating the semispinalis capitis muscle and the areas where they are concentrated were determined, the innervation map of the muscle was created. In this way, a muscle-nerve map was created as a guide for clinical applications.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Gözener Canbülbül, PhD(c), Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, Kavacık, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Robbins MS, Kuruvilla D, Blumenfeld A, Charleston L 4th, Sorrell M, Robertson CE, Grosberg BM, Bender SD, Napchan U, Ashkenazi A; Peripheral Nerve Blocks and Other Interventional Procedures Special Interest Section of the American Headache Society. Trigger point injections for headache disorders: expert consensus methodology and narrative review. Headache. 2014 Oct;54(9):1441-59. doi: 10.1111/head.12442. Epub 2014 Aug 28. PMID 25168295
- [Result] Rezasoltani A, Ahmadipoor A, Khademi-Kalantari K, Javanshir K. The sign of unilateral neck semispinalis capitis muscle atrophy in patients with chronic non-specific neck pain. J Back Musculoskelet Rehabil. 2012;25(1):67-72. doi: 10.3233/BMR-2012-0303. PMID 22398268
- [Result] Kaya B, Apaydin N, Loukas M, Tubbs RS. The topographic anatomy of the masseteric nerve: A cadaveric study with an emphasis on the effective zone of botulinum toxin A injections in masseter. J Plast Reconstr Aesthet Surg. 2014 Dec;67(12):1663-8. doi: 10.1016/j.bjps.2014.07.043. Epub 2014 Aug 7. PMID 25175271
- [Result] Takebe K, Vitti M, Basmajian JV. The functions of semispinalis capitis and splenius capitis muscles: an electromyographic study. Anat Rec. 1974 Aug;179(4):477-80. doi: 10.1002/ar.1091790407. No abstract available. PMID 4842939
- [Result] Elliott JM, O'Leary SP, Cagnie B, Durbridge G, Danneels L, Jull G. Craniocervical orientation affects muscle activation when exercising the cervical extensors in healthy subjects. Arch Phys Med Rehabil. 2010 Sep;91(9):1418-22. doi: 10.1016/j.apmr.2010.05.014. PMID 20801261